CLINICAL TRIAL: NCT07342569
Title: The WeACT Program for Family Caregivers of People Living With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Areum Han, Associate Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY009455; 7R21AG085254-02 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Depression; Caregivers; Dementia
Keywords: acceptance and commitment therapy; Internet-Based Intervention; caregivers; dementia; depressive symptoms; feasibility; usability; web-based intervention; mixed methods; Pilot Study
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and commitment therapy (ACT) group (Experimental): The ACT group will complete the WeACT program, a self-paced, web-based ACT program that includes six weekly online modules and a daily practice section.
  Interventions: Behavioral: WeACT

INTERVENTIONS:
Behavioral: WeACT — WeACT includes six self-paced weekly ACT modules and a tailored daily practice component. Each weekly module includes ACT skills training materials. The daily practice section provides brief, in-the-moment ACT skill coaching based on participants' current self-ratings.

SUMMARY:
The goal of this clinical trial is to learn whether WeACT, a self-paced, web-based program, is feasible and helpful for adult family caregivers of a relative living with dementia. WeACT is based on acceptance and commitment therapy (ACT), which teaches skills to handle difficult thoughts and feelings and take steps toward what matters most.

The main questions this study aims to answer are:

* Can caregivers complete WeACT as planned?
* Do caregivers show improvements in mental health and coping after using WeACT?
* What are caregivers' experiences with the program, and what suggestions do they have to improve it?

Participants will:

* Complete six self-paced weekly online modules and use the daily practice section during the program.
* Complete online questionnaires before starting and after completing the program.
* Take part in one online interview about their experience.

DETAILED DESCRIPTION:
Family caregivers of people living with dementia often experience psychological distress (such as depressive symptoms and stress) and face practical barriers to accessing support. This study will evaluate WeACT, a research-developed, self-paced, web-based acceptance and commitment therapy (ACT) skills program designed to support caregivers' mental health outcomes in a scalable format. This is a one-group, pretest-posttest mixed-methods pilot study conducted fully online. All enrolled participants will receive access to the WeACT program. The study will assess feasibility and user experience and will explore pre-to-post changes in caregiver mental health outcomes and ACT-related processes. WeACT includes six self-paced weekly ACT modules and a tailored daily practice component. Each weekly module includes ACT skills training materials. The daily practice section provides brief, in-the-moment ACT skill coaching based on participants' current self-ratings. Recruitment will occur by distributing a study flyer across the United States. Interested individuals will contact the study team and complete an online eligibility screening survey. Eligible individuals will complete electronic informed consent and then complete pretest questionnaires online. After completing baseline procedures, participants will receive program access and study-specific login credentials. Participants will be encouraged to complete one module per week and to use the daily practice section regularly during the intervention period. After completing the program modules, participants will complete posttest questionnaires online and participate in a one-time individual interview. Interviews will be conducted and recorded using the HIPAA-compliant version of Microsoft Teams. Feasibility will be evaluated using recruitment, retention, and adherence indicators and by documenting reasons for ineligibility and dropout. The program will also capture engagement and in-program response data. Pretest and posttest questionnaires will be used to explore changes in caregiver mental health outcomes and ACT-related processes and to assess perceived feasibility, acceptability, appropriateness, and usability at posttest. Qualitative interviews will be used to understand participant experiences and identify recommendations to refine the program and study procedures. Analyses will focus on feasibility and descriptive characterization of engagement. Pre-to-post changes will be explored using paired statistical tests as appropriate. Daily practice data will be explored using multilevel modeling to estimate average change and individual variability over time. Interview data will be analyzed using thematic analysis to summarize common experiences and improvement suggestions. All data will be collected electronically using university-approved secure platforms (Qualtrics, the WeACT program hosted on the secure USF Microsoft Azure environment, and HIPAA-compliant Microsoft Teams). WeACT is not publicly available and is accessible only to enrolled participants. Participants will use study-specific login credentials. Identifying information will be collected only as needed for study operations (e.g., communication and compensation) and stored separately from research data. Study data will be stored in secure, access-controlled USF systems (including USF Box), with access restricted to authorized study personnel. Only de-identified, aggregate results will be used for dissemination.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling adults (aged 18 years or older) who have primary caregiving responsibilities for a relative diagnosed with dementia;
2. Present mild to moderate depressive symptoms, as measured by the Patient Health Questionnaire-9 (PHQ-9), with scores between 5 and 14; and
3. Have access to a web-enabled device (i.e., a smartphone, tablet, laptop, or desktop) with internet access

Exclusion Criteria:

1. Cognitive, physical, or sensory impairments, or language barriers (non-English communicator) that might impede study participation;
2. Present moderately severe to severe depressive symptoms, defined as PHQ-9 scores between 15 and 27;
3. Have previously participated in a research study that involved an ACT program;
4. Have suicidal intent or a suicide attempt within the past six months;
5. Are currently participating in another caregiver study; or
6. Have experienced more than three hospitalizations (of either the family caregiver or the relative with dementia) within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | During the recruitment period (up to approximately 6 months)
  Enrollment rate will be defined as the number of individuals who consent and complete baseline divided by the number eligible and invited.
Retention (post-intervention assessment completion) | Baseline through post-intervention (approximately 6-8 weeks)
  Retention will be defined as the proportion of enrolled participants who complete the post-intervention assessment.
Core module completion (adherence) | During program participation (~6-8 weeks)
  Adherence will be defined as completion of the core modules (range 0-6 modules).

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | Post-intervention (~6-8 weeks)
  4-item acceptability rating (5-point Likert-type responses; 1 = completely disagree to 5 = completely agree).
Intervention Appropriateness Measure | Post-intervention (~6-8 weeks)
  4-item appropriateness rating (5-point Likert-type responses; 1 = completely disagree to 5 = completely agree).
Feasibility of Intervention Measure | Post-intervention (~6-8 weeks)
  4-item perceived feasibility rating (5-point Likert-type responses; 1 = completely disagree to 5 = completely agree).
System Usability Scale (SUS) | Post-intervention (approximately 6-8 weeks)
  10-item usability measure (5-point Likert); interpreted using common benchmarks (e.g., ~68 average; ≥70 acceptable).
Change in Patient Health Questionnaire-9 (PHQ-9) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  PHQ-9 is a nine-item self-report questionnaire assessing depressive symptoms over the past two weeks, rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in Generalized Anxiety Disorder -7 (GAD-7) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  GAD-7 is a seven-item self-report questionnaire assessing anxiety symptoms over the past two weeks, rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with higher scores reflecting greater anxiety symptoms.
Change in Perceived Stress Scale-10 (PSS-10) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  PSS-10 is a 10-item questionnaire assessing stress on a scale of 0 to 4. Scores range from 0 to 40. Higher scores indicate greater stress.
Change in World Health Organization Quality of Life-BREF (WHOQOL-BREF) - Psychological Health Subscale scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  WHOQOL-BREF - Psychological Health Subscale has 6 items measuring psychological quality of life on a scale of 1 to 5. The total scores range from 6 to 30. Higher scores denote a higher quality of life in terms of psychological health.
Change in Zarit Burden Interview (ZBI) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  ZBI is a 12-item self-report questionnaire assessing caregiver burden on a scale of 0 to 4. The total scores range from 0 to 48. Higher scores indicate higher burden levels.
Change in Marwit-Meuser Caregiver Grief Inventory-Brief Form (MM-CGI-BF) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  MM-CGI-BF is a six-item self-report questionnaire that assesses pre-death grief in caregivers of people with dementia, rated on a scale from 1 to 5. Scores range from 6 to 30, with higher scores indicating greater grief.
Change in Caregiver Guilt Questionnaire (CGQ) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  CGQ is a 22-item self-report measure that assesses feelings of guilt in caregivers, rated on a scale from 0 to 4. Scores range from 0 to 88, with higher scores indicating greater levels of guilt.
Change in Acceptance and Action Questionnaire-II (AAQ-II) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  AAQ-II is a 7-item self-report questionnaire measuring psychological inflexibility on a scale of 1 to 7. The total scores range from 7 to 49, and higher scores indicate poor psychological flexibility.
Change in Cognitive Fusion Questionnaire-7 (CFQ-7) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  CFQ-7 is a 7-item self-report questionnaire measuring cognitive fusion on a scale of 1 to 7. The total scores range from 7 to 49, and higher scores indicate a higher degree of cognitive fusion.
Change in Engaged Living Scale-9 (ELS-9) scores from baseline to post-intervention | Baseline to post-intervention (approximately 6-8 weeks)
  ELS-9 is a 9-item self-assessment instrument that measures clarity and engagement with personal values and life fulfillment on a scale of 1 to 5. The total scores range from 9 to 45, and higher scores indicate increased clarity and engagement with personal values.

OTHER OUTCOMES:
User experiences (Semi-structured individual interviews) | Post-intervention (approximately 6-8 weeks)
  Individual interviews (~40 minutes) will be conducted via videoconference to explore user experiences (e.g., perceived impact, usability/access, and suggestions for improvement).
In-app daily ACT skills practice use | During program participation (~6-8 weeks)
  Number of self-initiated, tailored ACT daily practices completed per participant (log-based).

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No